CLINICAL TRIAL: NCT02631590
Title: Phase II Study of Copanlisib (BAY 80-6946) in Combination With Gemcitabine and Cisplatin in Advanced Cholangiocarcinoma
Brief Title: Copanlisib (BAY 80-6946) in Combination With Gemcitabine and Cisplatin in Advanced Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18435
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Biliary Carcinoma; Gall Bladder Carcinoma; Cholangiocarcinoma; Gastrointestinal Tumor
Keywords: intra-hepatic biliary system; extra-hepatic biliary system; gall bladder; advanced biliary cancer; unresectable; locally advanced; metastatic disease
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma; Digestive System Neoplasms; Neoplasm Metastasis | interventions — Cisplatin; Gemcitabine; copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Therapy (Experimental): Treatment Plan: Cisplatin (25 mg/m^2 ) + Gemcitabine (1000 mg/m^2) + copanlisib (60 mg) on days 1 and 8 with day 15 off to be administered on an every 21-days schedule.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Copanlisib

INTERVENTIONS:
Drug: Cisplatin — Cisplatin administered once as intravenous (IV) infusion over 60 minutes. Treatment is on Days 1 and 8 every 21 days.
  Other Names: Platinol
Drug: Gemcitabine — Gemcitabine administered as 30-min IV infusion. Treatment is on Days 1 and 8 every 21 days.
  Other Names: Gemzar
Drug: Copanlisib — Experimental Drug: Copanlisib administered as an IV over 60-minutes beginning 1 hour after completing gemcitabine infusion. Treatment is on Days 1 and 8 every 21 days.
  Other Names: BAY 80-6946

SUMMARY:
The purpose of this study is to see if an experimental drug, called copanlisib is effective and safe in treating adult participants with cholangiocarcinoma, when used in combination with gemcitabine and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically documented carcinoma primary to the intra- or extra-hepatic biliary system or gall bladder with clinical and/or radiologic evidence of unresectable, locally advanced or metastatic disease. Patients with ampullary carcinoma are not eligible.
* Must not have received any systemic chemotherapy for advanced biliary cancer.
* Patients who received adjuvant chemotherapy plus or minus radiation and had evidence of disease recurrence within 6 months of completion of the adjuvant treatment are not eligible. If patients received adjuvant treatment and had disease recurrence after 6 months, patients will be eligible.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Assessment of 0 or 1.
* Must have radiographic measurable disease.
* Life expectancy of at least 12 weeks (3 months).
* For patients who have received prior radiation, cryotherapy, radiofrequency ablation, therasphere, ethanol injection, transarterial chemoembolization (TACE) or photodynamic therapy, the following criteria must be met: 28 days have elapsed since that therapy; Lesions that have not been treated with local therapy must be present and measureable.
* Adequate bone marrow, liver and liver function.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Men and women of childbearing potential must agree to use adequate contraception beginning at the signing of the Informed Consent Form (ICF) until at least 3 months after the last dose of study drug.
* Must be able to swallow and retain oral medication.
* Availability of archival tumor tissue for biomarkers analysis (minimum of 10 unstained slides are optional). Specimen from primary site will be allowed.

Exclusion Criteria:

* Previous or concurrent cancer within 3 years prior to treatment start except for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Congestive heart failure > New York Heart Association (NYHA) class 2.
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months).
* Myocardial infarction less than 6 months before study enrollment
* Uncontrolled hypertension (blood pressure ≥ 150/90 mmHg despite optimal medical management).
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before enrollment.
* Non-healing wound, ulcer, or bone fracture.
* Active clinically serious infections (> Common Terminology Criteria for Adverse Events (CTCAE) grade 2).
* Known history of human immunodeficiency virus (HIV) infection.
* Known active Hepatitis B or C.
* A seizure disorder requiring medication.
* Evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks of start of study enrollment.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Known hypersensitivity to any of the test drugs, test drug classes, or excipients in the formulation.
* History or concurrent condition of interstitial lung disease of any grade or severely impaired pulmonary function.
* Unresolved toxicity higher than CTCAE grade 1 attributed to any prior therapy/procedure excluding alopecia.
* HbA1c >8.5% or fasting plasma glucose > 160 mg/dL at screening.
* Concurrent diagnosis of pheochromocytoma.
* Women who are pregnant or breast feeding.
* Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his/her compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2021-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Kim, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Tan ES, Cao B, Kim J, Al-Toubah TE, Mehta R, Centeno BA, Kim RD. Phase 2 study of copanlisib in combination with gemcitabine and cisplatin in advanced biliary tract cancers. Cancer. 2021 Apr 15;127(8):1293-1300. doi: 10.1002/cncr.33364. Epub 2020 Dec 8. PMID 33289918
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Therapy
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants that received at least one dose of study drug
Arm/Group | Combination Therapy
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS at six months. Response and progression will be evaluated using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1). PFS will be calculated from study entry to documented disease progression, death from any cause, or date of last follow-up, whichever comes first. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression.)
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 24
months | 6.2 [2.9 to 10.1]

2. Secondary Outcome: Response Rate
Description: Complete Response + Partial Response according to RECIST 1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 24 months
Population: Number of participants evaluable for response
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 19
percentage of participants
  Partial Response | 31.6
  Stable Disease | 57.9

3. Secondary Outcome: Overall Survival (OS)
Description: The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 24
months | 13.7 [6.8 to 18.0]

ADVERSE EVENTS:
Time Frame: All adverse events collected from start of study drug to 4 weeks after end of treatment, 2 years 3 months.
Arm/Group | Combination Therapy
All-Cause Mortality (participants affected / at risk) | 18/24
Serious Adverse Events (participants affected / at risk) | 12/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=24)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Hepatic infection (Hepatobiliary disorders) | 1 (2)
Infections and Infestations - Other (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=24)
Nausea (Gastrointestinal disorders) | 12 (22)
Diarrhea (Gastrointestinal disorders) | 11 (12)
Abdominal Pain (Gastrointestinal disorders) | 10 (13)
Constipation (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 6 (13)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 17 (27)
Fever (General disorders) | 8 (24)
Edema limbs (General disorders) | 5 (6)
Chills (General disorders) | 4 (7)
Pain (General disorders) | 4 (4)
Infusion related reaction (General disorders) | 3 (4)
Non-cardiac chest pain (General disorders) | 3 (6)
General disorders and administration site conditions -Other (General disorders) | 2 (2)
Gait disturbance (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 18 (66)
Platelet count decreased (Investigations) | 18 (45)
White blood cell decreased (Investigations) | 17 (72)
Neutrophil count decreased (Investigations) | 16 (62)
Lipase increased (Investigations) | 11 (33)
Alanine aminotransferase increased (Investigations) | 10 (21)
Weight loss (Investigations) | 6 (15)
Aspartate aminotransferase increased (Investigations) | 5 (15)
Serum amylase increased (Investigations) | 5 (9)
Alkaline phosphatase increased (Investigations) | 4 (8)
Creatinine increased (Investigations) | 4 (5)
Blood bilirubin increased (Investigations) | 3 (6)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Blood antidiuretic hormone abnormal (Investigations) | 1 (1)
Investigations - Other (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (43)
Anorexia (Metabolism and nutrition disorders) | 11 (14)
Hyponatremia (Metabolism and nutrition disorders) | 7 (10)
Dehydration (Metabolism and nutrition disorders) | 6 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 16 (56)
Hypertension (Vascular disorders) | 15 (54)
Hypotension (Vascular disorders) | 6 (8)
Thromboembolic event (Vascular disorders) | 4 (9)
Phlebitis (Vascular disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorders - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (5)
Headache (Nervous system disorders) | 1 (1)
Parathesia (Nervous system disorders) | 1 (2)
Sepsis (Infections and infestations) | 3 (3)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (4)
Infections and infestations - Other (Infections and infestations) | 2 (5)
Gallbladder infection (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (2)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1)
Venous injury (Injury, poisoning and procedural complications) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT02631590/Prot_SAP_000.pdf